CLINICAL TRIAL: NCT06648564
Title: 20-25 Year Follow-Up After Surgical Treatment of Peri-Implantitis Using a Bone Substitute with or Without a Resorbable Membrane: a Longitudinal Study
Brief Title: 20-25 Year Follow-Up on Regenerative Bone Procedures for Peri-Implantitis
Acronym: periimpl20y
Status: Enrolling by invitation | Type: Observational
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Viveca Wallin Bengtsson, phD, Kristianstad University
Other Study IDs: P-i regenerative surg 20-25 y
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peri-implantitis
Keywords: peri-implantitis; regenerative surgery; long time follow-up
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Bone regenerativ surgery with a bone graft material (Algipore) and a resorbable membrane (Osseoquest)
  Interventions: Procedure: Bone regenerative surgery with a bone graft substitute and a resorbable membrane
- Group 2: Bone regenerativ surgery with a bone graft material (Algipore)

INTERVENTIONS:
Procedure: Bone regenerative surgery with a bone graft substitute and a resorbable membrane — Dental implants with a diagnosis peri-implantitis were treated with regenerative surgery.
  Other Names: Bone regenerative surgery with a bone graft substitute
  Groups: Group 1

SUMMARY:
The goal of this 20-25-year observational study is to investigate the outcomes of bone regenerative surgery in peri-implantitis. Two different techniques will be compared: surgery with a bone substitute alone and surgery with a bone substitute combined with a membrane, to determine their effectiveness and assess whether one is more effective than the other. The intention of this observational study is to learn more about the long-term effects of bone regenerative surgery in patients with peri-implantitis.

Patients will be called in for a clinical and radiographic examination of the surgically treated implant(s). Probing pocket depths, presence of pus, bleeding around the implant (s) and a radiograph of the implant (s).

To be able to compare with the 1, 3, 5 and 10 year measurements.

DETAILED DESCRIPTION:
The aim of this 20-25 year observational follow-up study is to investigate the outcomes of bone regenerative surgery in peri-implantitis. The study compares two approaches: Group 1: surgery with a bone substitute alone (Algipore) and Group 2: surgery with a bone substitute (Algipore) combined with a membrane (Osseoquest). Both groups received systemic antibiotics-Amoxicillin 375 mg three times a day combined with Metronidazole 400 mg twice a day for 10 days, starting the day before surgery.

The objective of this observational study is to gain insights into the long-term effects of bone regenerative surgery in patients with peri-implantitis and to determine if there is a difference.

The patients were enrolled in a strict maintenance program with supportive therapy every third months with a yearly evaluation.

In this study, patients will examined of the surgically treated implant(s) after 20-25 years. The examination will include a clinical assessment, measuring probing pocket depths at each implant to the nearest millimeter using a standardized probing force of 0.25 N (Hawe-Click Probe, Kerr Hawe SA Bioggio, Switzerland). The prevalence of pus, full-mouth bleeding on probing, and bleeding grades will be recorded around the implant(s) at four sites per tooth and implant(s) as follows: 0 = no bleeding, 1 = point of bleeding, 2 = line of bleeding, and 3 = drop of bleeding. The plaque index will be defined as either visible or not visible at the implant site using an erythrosine dye (TopDent Lifco Dental AB, Enköping, Sweden). All clinical assessments will be performed by the same periodontist (AMRJ).

Data from the clinical treatment were registered in patient records. In parallel, clinical data were documented in a study protocol and saved in a safe in accordance with standard operation procedure at the clinic.The protocol with medical records were not opened until the study was completed and only by authorized persons with access to the data in the study such as, principal investigator and statisticians.

In accordance with an international working group diagnosis of peri-implantitis should include pocket depth, bleeding, and bone loss (X-ray). Thus, in this study the primary outcomes are radiographic evidence of bone fill and changes in probing depths at implants treated.

Parametric tests (independent t-tests, equal variance not assumed), and non-parametric tests (Mann-Whitney U-test, Wilcoxon test) will be performed to assess differences over time and between groups. Statistical significance will be declared at p <0.05. The Kolmogorov- Smirnov test will be used to define if the data presented with normal distribution or not. The SPSS PASW 29.0 statistical software (SPSS Inc., Chicago, IL, USA) for Apple computer will be used in the analysis.

Patients that will participate in the study will consecutively be given an ID code. and data will be registered in the ordinary patient journal. The code list will be placed in a locked up space, at the clinic.

All patients will be given oral and written information about the study and will sign a written informed consent. The patients will be informed that they could drop off when ever they want without any explanations. The ethical board approved the study.

ELIGIBILITY:
Inclusion Criteria:

* An implant demonstrating a progressive bone loss of ≥3 threads (≥1.8 mm) following the first year of healing
* A vertical component needed to be present at the surgical intervention in order to justify the use of a bone augmentation procedure.
* Bleeding on probing and/or suppuration should also be present

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with at least one dental implant with peri-implantitis
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone fill | Ten years after surgical regenerative boneprocedures
  Radiographic bone fill measured mesial and distal at the implant on an intra oral radiograph. Measurements will be performed by a blinded radiologist.

SECONDARY OUTCOMES:
Probing pocket depths changes | Ten years after surgical regenerative boneprocedures
  Changes in probing pocket depth at the implant measured on 4 surfaces

OTHER OUTCOMES:
Bleeding | Ten years after surgical regenerative boneprocedures
  Bleeding on probing measured at the implant on 4 sites.
Graded bleeding | Ten years after surgical regenerative boneprocedures
  Graded bleeding measured at the implant on 4 sites as: 0 = no bleeding, 1 = point of bleeding, 2 = line of bleeding, and 3 = drop of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: AM R Jansaker, Ass.Prof., Study Director — Malmö University; Stefan Renvert, Prof., Study Chair — Kristianstad University
Locations (1):
- Kristianstad Univeristy, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
May be shared upon request

REFERENCES:
- [Background] Roos-Jansaker AM, Persson GR, Lindahl C, Renvert S. Surgical treatment of peri-implantitis using a bone substitute with or without a resorbable membrane: a 5-year follow-up. J Clin Periodontol. 2014 Nov;41(11):1108-14. doi: 10.1111/jcpe.12308. Epub 2014 Oct 17. PMID 25195613
- [Background] Roos-Jansaker AM, Lindahl C, Persson GR, Renvert S. Long-term stability of surgical bone regenerative procedures of peri-implantitis lesions in a prospective case-control study over 3 years. J Clin Periodontol. 2011 Jun;38(6):590-7. doi: 10.1111/j.1600-051X.2011.01729.x. Epub 2011 Apr 13. PMID 21488935
- [Background] Roos-Jansaker AM, Renvert H, Lindahl C, Renvert S. Surgical treatment of peri-implantitis using a bone substitute with or without a resorbable membrane: a prospective cohort study. J Clin Periodontol. 2007 Jul;34(7):625-32. doi: 10.1111/j.1600-051X.2007.01102.x. PMID 17555414